CLINICAL TRIAL: NCT02575911
Title: Accuracy of LASIK Flaps Created With the LenSx® Femtosecond Laser - A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTJ121-P001
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-04

CONDITIONS: Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- LenSx (Experimental): LASIK surgery in both eyes using LenSx® Femtosecond Laser System
  Interventions: Device: Femtosecond Laser System; Procedure: LASIK surgery

INTERVENTIONS:
Device: Femtosecond Laser System — Used for the creation of a corneal flap in patients undergoing LASIK surgery
  Other Names: LenSx®
Procedure: LASIK surgery

SUMMARY:
The purpose of this study is to evaluate the thickness accuracy of Laser-assisted in situ keratomileusis (LASIK) flaps created with the LenSx® Laser.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with myopia or hyperopia and eligible for femtosecond laser initiated LASIK surgery;
* Best corrected visual acuity (BCVA) correctable to at least 20/25 in each eye;
* If contact lens wearer, willing to discontinue contact lens wear prior to screening procedures;
* Willing and able to return for ALL scheduled follow-up examinations;
* Willing and able to provide written informed consent;
* Eligible for bilateral LASIK procedures to be done on the same day;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Previous corneal surgery, corneal lesions that will impede laser treatment, corneal edema, hypotony, glaucoma, existing corneal implant, or keratoconus;
* Known sensitivity to planned study concomitant medications;
* Participation in any other ophthalmic drug or device clinical study for 30 days prior to or during the time of participation in this study;
* Irregular astigmatism, based on the Investigator's judgement;
* Pregnant, lactating or planning to become pregnant during the course of the study;
* Other protocol-specified exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2016-04-09 (Actual); Study Completion 2016-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Manager, GCRA, Study Director — Alcon, A Novartis Division
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 2 sites located in the US.
Pre-assignment Details: Of the 34 enrolled, 4 participants were exited as screen failures prior to surgery. This reporting group includes all treated participants (30).
Period: Overall Study
Arm/Group | LenSx
Started | 30
Completed | 29
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all participants/eyes exposed to the device during the study (Safety Analysis Set).
Arm/Group | LenSx
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Flap Thickness Accuracy Within the Central Zone at Month 3 Postoperative
Description: Flap thickness was assessed by optical coherence tomography (OCT) and averaged from 3 separate scans. Flap thickness accuracy was defined as the mean difference between the achieved and desired (desired subtracted from achieved) flap thickness. A positive number represents a postoperative flap thickness that is thicker than the expected flap thickness and vice versa for a negative number. Each eye contributed separately to the analysis.
Time Frame: Month 3 postoperative
Population: This analysis population includes the number of eyes treated with surgery and data available.
Measure: Mean (Standard Deviation); unit: micrometers
Units Other Than Participants: Eyes
Arm/Group | LenSx
Number analyzed (Participants) | 29
Number analyzed (Eyes) | 58
micrometers | 125.8 (4.8)

2. Secondary Outcome: Flap Thickness Accuracy Within the Central Zone at Month 1 Postoperative
Description: Flap thickness was assessed by OCT and averaged from 3 separate scans. Flap thickness accuracy was defined as the mean difference between the achieved and desired (desired subtracted from achieved) flap thickness. A positive number represents a postoperative flap thickness that is thicker than the expected flap thickness and vice versa for a negative number. Each eye contributed separately to the analysis.
Time Frame: Month 1 postoperative
Population: This analysis population includes the number of eyes treated with surgery and data available.
Measure: Mean (Standard Deviation); unit: micrometers
Units Other Than Participants: Eyes
Arm/Group | LenSx
Number analyzed (Participants) | 29
Number analyzed (Eyes) | 58
micrometers | 127.8 (3.7)

3. Secondary Outcome: Flap Thickness Precision Within the Central Zone at Month 1 and Month 3 Postoperative
Description: Flap thickness was assessed by OCT and averaged from 3 separate scans. Flap thickness precision (variability of the achieved flap thickness) was defined as the standard deviation of the flap thickness measurement. Each eye contributed separately to the analysis.
Time Frame: Month 1, Month 3 postoperative
Population: This analysis population includes the number of eyes treated with surgery and data available.
Measure: Mean (Standard Deviation); unit: micrometers
Units Other Than Participants: Eyes
Arm/Group | LenSx
Number analyzed (Participants) | 29
Number analyzed (Eyes) | 58
micrometers
  Month 1 postoperative | 127.8 (3.7)
  Month 3 postoperative | 125.8 (4.8)

4. Secondary Outcome: Ease of Flap Dissection at Day 0, Operative Day
Description: Ease of flap dissection (ease of lifting the flap during surgery) was assessed on a scale from 0 to 5 where 0 = Unable to lift flap and 5 = Able to lift flap without any resistance using blunt instrument. Each eye contributed separately to the analysis.
Time Frame: Day 0, operative day
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | LenSx
Number analyzed (Participants) | 30
Number analyzed (Eyes) | 60
units on a scale | 4.7 (0.5)

5. Secondary Outcome: Stromal Bed Quality at Day 0, Operative Day
Description: Stromal bed quality was assessed by the investigator on a roughness scale from 0 to 5 where 0 = Very rough surface and 5 = Very smooth surface. Each eye contributed separately to the analysis.
Time Frame: Day 0, operative day
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | LenSx
Number analyzed (Participants) | 30
Number analyzed (Eyes) | 60
units on a scale | 5.0 (0.0)

6. Secondary Outcome: Opaque Bubble Layer (OBL) at Day 0, Operative Day
Description: Opaque bubble layer was assessed by the investigator during the surgery on a scale from 0 to 5 where 0 = No OBL and 5 = 100% OBL in the stromal bed area. Each eye contributed separately to the analysis.
Time Frame: Day 0, operative day
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | LenSx
Number analyzed (Participants) | 30
Number analyzed (Eyes) | 60
units on a scale | 0.3 (0.4)

7. Secondary Outcome: Uncorrected Distance Visual Acuity (UCDVA) at Month 1 and Month 3 Postoperative
Description: UCDVA (measurement of uncorrected (without spectacles or other visual corrective devices) distance visual acuity) was assessed at a distance of 6 meters or 20 feet using a standard Snellen eye chart, both monocularly and binocularly, and reported categorically as a percentage of eyes analyzed.
Time Frame: Month 1, Month 3 postoperative
Population: This analysis population includes the number of eyes treated with surgery and data available.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Groups:
- LenSx - Month 1 Postoperative: LASIK surgery in both eyes using LenSx® Femtosecond Laser System, 1 month post-operative
- LenSx - Month 3 Postoperative: LASIK surgery in both eyes using LenSx® Femtosecond Laser System, 3 months post-operative
Arm/Group | LenSx - Month 1 Postoperative | LenSx - Month 3 Postoperative
Number analyzed (Participants) | 29 | 29
Number analyzed (Eyes) | 58 | 58
percentage of eyes
  ≤ 20/15 | 0.0 | 0.0
  20/20 | 81.0 | 84.5
  20/25 | 8.6 | 6.9
  20/30 | 5.2 | 3.4
  20/40 | 0.0 | 3.4
  >20/40 | 5.2 | 1.7

8. Secondary Outcome: Best Corrected Distance Visual Acuity (BCDVA) by Visit
Description: BCDVA (measurement with the participant's best spectacle correction) was assessed at a distance of 6 meters or 20 feet using a standard Snellen eye chart, both monocularly and binocularly, and reported categorically as a percentage of eyes analyzed.
Time Frame: Baseline, Month 1, Month 3 postoperative
Population: This analysis population includes total number of eyes in specified category at visit.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Groups:
- Baseline: Prior to LASIK surgery
Arm/Group | Baseline | LenSx - Month 1 Postoperative | LenSx - Month 3 Postoperative
Number analyzed (Participants) | 30 | 29 | 29
Number analyzed (Eyes) | 60 | 58 | 58
percentage of eyes
  ≤ 20/15 | 0.0 | 1.7 | 0.0
  20/20 | 91.7 | 91.4 | 98.3
  20/25 | 8.3 | 3.4 | 1.7
  20/30 | 0.0 | 0.0 | 0.0
  20/40 | 0.0 | 1.7 | 0.0
  >20/40 | 0.0 | 1.7 | 0.0

9. Secondary Outcome: Manifest Refraction Spherical Equivalent (MRSE)
Description: The participant was manually refracted to his/her best correction using a phoropter and standard Snellen eye charts. Each eye contributed separately to the analysis.
Time Frame: Baseline, Month 1, Month 3 postoperative
Population: This analysis population includes number of eyes in specified category.
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: Eyes
Arm/Group | LenSx
Number analyzed (Participants) | 30
Number analyzed (Eyes) | 60
diopter
  Baseline | -2.846 (2.090)
  Month 1 postoperative: number analyzed (Eyes) | 58
  Month 1 postoperative | -0.194 (0.329)
  Month 3 postoperative: number analyzed (Eyes) | 58
  Month 3 postoperative | -0.166 (0.307)

10. Secondary Outcome: Prediction Error Between Target Versus Achieved Refraction at One and Three Months Post-op
Description: Prediction error was summarized as a percentage of eyes within 0.5 D and 1.0 D of target at one and three months postoperative
Time Frame: Month 1, Month 3 postoperative
Population: This analysis population includes the number of eyes treated with surgery and data available at the specified time point.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Groups:
- LenSx - 1 Month Postoperative: LASIK surgery in both eyes using LenSx® Femtosecond Laser System, 1 month post-operative
- LenSx - 3 Months Postoperative: LASIK surgery in both eyes using LenSx® Femtosecond Laser System, 3 months post-operative
Arm/Group | LenSx - 1 Month Postoperative | LenSx - 3 Months Postoperative
Number analyzed (Participants) | 29 | 29
Number analyzed (Eyes) | 58 | 58
percentage of eyes
  0.5 diopter (D) | 93.1 | 91.4
  1.0 D | 98.3 | 100.0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of participation in the study (up to 5 months). AEs are reported as pre-treatment and treatment-emergent. "At Risk" population for ocular AEs is included with unit of "eyes."
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the medical device.
Groups:
- Pre-treatment: All who consented to participate in the study prior to the initiation of study treatment
- LenSx: All subjects treated with LASIK surgery in both eyes using LenSx® Femtosecond Laser System
Arm/Group | Pre-treatment | LenSx
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/68 | 1/60
Other Adverse Events (participants affected / at risk) | 0/68 | 7/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-treatment (N=68) | LenSx (N=60)
Corneal striae (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-treatment (N=68) | LenSx (N=60)
Punctate keratitis (Eye disorders) | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.